CLINICAL TRIAL: NCT07392372
Title: A Phase I First-in-human Clinical Trial to Evaluate the Safety, Pharmacokinetics, and Antiviral Activity of the Broadly Neutralizing Antibody BNT351 in Adults Living Without and With HIV
Brief Title: A Clinical Trial Investigating the Safety and Biological Activity of the Antibody BNT351 in Adults Living Without and With HIV
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNT351-01; 2025-523846-29-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: HIV -1 Infection
Keywords: HIV-1; Treatment of HIV-1 infection; Antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A - Cohort A1 (Experimental): PLWOH will be randomized to BNT351 (at a protocol defined dose level) or placebo (2:1)
  Interventions: Drug: BNT351; Drug: Placebo
- Part A - Cohort A2 (Experimental): PLWOH will be randomized to BNT351 (at a protocol defined dose level) or placebo (3:1)
  Interventions: Drug: BNT351; Drug: Placebo
- Part A - Cohort A3 (Experimental): PLWOH will be randomized to BNT351 (at a protocol defined dose level) or placebo (3:1)
  Interventions: Drug: BNT351; Drug: Placebo
- Part A - Cohort A4 (Experimental): PLWOH will be randomized to BNT351 (at a protocol defined dose level) or placebo (3:1)
  Interventions: Drug: BNT351; Drug: Placebo
- Part B - Cohort B1 (Experimental): PLWH will receive BNT351 at a protocol-defined dose level. cART will start 56 days post-BNT351 dosing or earlier.
  Interventions: Drug: BNT351

INTERVENTIONS:
Drug: BNT351 — IV infusion
  Arms: Part A - Cohort A2; Part A - Cohort A3; Part A - Cohort A4; Part B - Cohort B1
Drug: Placebo — IV infusion
  Arms: Part A - Cohort A2; Part A - Cohort A3; Part A - Cohort A4
Drug: BNT351 — SC injection
  Arms: Part A - Cohort A1
Drug: Placebo — SC injection
  Arms: Part A - Cohort A1

SUMMARY:
This study will test the safety and blood levels of the antibody BNT351 in people living without and with human immunodeficiency virus (HIV). This study will also test the anti-viral activity of BNT351 in people living with HIV (PLWH) with detectable virus levels.

The main goals of this study are:

* To learn about the safety of BNT351 and check for side effects.
* To measure the amount of BNT351 antibody in blood over time.
* To test the amount of HIV in the blood at different times after treatment with BNT351 in people living with HIV.

DETAILED DESCRIPTION:
The study will consist of two parts (Parts A and B).

Part A will be a randomized, double-blind, placebo-controlled, single ascending dose, first-in-human study part. Part A will enroll people living without HIV (PLWOH). Four cohorts are planned in Part A (Cohorts A1, A2, A3, and A4). Cohort A1 will evaluate one dose of BNT351 administered subcutaneously (SC). Cohorts A2 to A4 will evaluate three different doses of BNT351 administered intravenously (IV). For each cohort, participants will be randomized to BNT351 or placebo.

Part B will be single-dose, open-label, proof-of concept study part. Part B will enroll PLWH. Part B comprises of a single cohort (Cohort B1) and will be non-randomized.

The study will start with recruitment into Part A. Part B will be opened after review of safety data from Part A.

In Part A, for each participant, there will be an ~4-week screening period, one dose of BNT351 or placebo, and an ~38-week follow-up period. In total, Part A will last up to ~42 weeks per participant.

In Part B, for each participant, there will be an ~4-week screening period, one dose of BNT351, and an up to 8-week observation period with HIV viral load assessments, after which combination antiretroviral therapy (cART) will be started. Overall, participants will be followed for ~38 weeks after IMP administration and in total, Part B will last up to ~42 weeks per participant.

ELIGIBILITY:
Key Inclusion Criteria

Part A:

* Are HIV-1 and HIV-2 negative at Visit 0.
* Starting at Visit 0 and continuously until the last planned visit in this study are individuals who:

  1. Are assessed by the investigator as having a low likelihood of acquiring HIV and are committed to avoiding behaviors associated with a higher likelihood of acquiring HIV until the End of Study Visit.
  2. Agree to discuss HIV disease risks;
  3. Agree to HIV acquisition risk reduction counseling;

Part B:

* Are HIV-1 positive and HIV-2 negative at Visit 0.
* Individuals who at Visit 0:

  1. Are cART-naïve individuals who were diagnosed with HIV-1 infection ≤12 months prior to screening, OR are individuals who have discontinued cART and who were diagnosed with HIV-1 infection ≤12 months prior to screening or ≤18 months if this is found to be acceptable after discussion on a case-by-case basis with the sponsor's medical monitor.
  2. If cART-experienced, have discontinued cART for at least 4 weeks before screening (if the individual was taking long-acting antiretroviral therapy [ART]), see the following bullet). For individuals who have discontinued cART: Are able to comply with study procedures and assessments in the investigator's judgment.
  3. Have never received lenacapavir and have not received other long-acting ARTs in the last 6 months (i.e., intramuscular cabotegravir, cabotegravir-rilpivirine).
  4. Have a CD4+ T cell count of ≥400 cells/µL and plasma HIV-1 RNA levels between 1,000-100,000 copies/mL at screening.
  5. Are willing to initiate cART at a protocol-defined timepoint (56 days post-dose, or earlier if meeting early cART start criteria or at investigator's discretion).
  6. Are willing to undergo HIV transmission risk reduction counseling and to maintain low-risk behavior to protect their partners.

Key Exclusion Criteria:

Part A:

* Have received an HIV vaccination or HIV broadly neutralizing antibody in another clinical study.
* Have a known or suspected impairment/alteration of immune function or immunodeficiency, including receipt of any immunostimulant, immunomodulator, immunosuppressive medication, immunoglobulin, blood product, or oral or parenteral steroid within 60 days prior to Day 1 or planned administration during the study. The following exception applies: Use of inhaled, intranasal, topical, or locally injected corticosteroids (e.g., intraarticular or intrabursal administration) is allowed.
* Have a history of generalized urticaria or angioedema, or of allergy, anaphylaxis, hypersensitivity or intolerance to a human or humanized antibody or to BNT351 excipients.

Part B:

* Have received an HIV vaccination or HIV broadly neutralizing antibody in another clinical study.
* Are receiving ongoing therapy for Mycobacterium tuberculosis infection.
* Have a history of opportunistic infections/AIDS-defining illnesses as defined in the protocol.
* Have a history of multi-class drug resistant HIV-1 infection defined as resistance to three or more classes of HIV drugs.
* Have a history of malignancy within 5 years before screening. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or a malignancy which is considered in the investigator's judgment to have minimal risk of recurrence. Any malignancy that is an AIDS-defining illness (as defined in the protocol) is exclusionary regardless of the perceived risk of recurrence.
* Have a known or suspected impairment/alteration of immune function or immunodeficiency (except for HIV infection), including receipt of any immunostimulant, immunomodulator, immunosuppressive medication, immunoglobulin, blood product, or oral or parenteral steroid within 60 days prior to Day 1 or planned administration during the study. The following exception applies: Use of inhaled, intranasal, topical, or locally injected corticosteroids (e.g., intraarticular or intrabursal administration) is allowed.
* Have a history of generalized urticaria or angioedema, or of allergy, anaphylaxis, hypersensitivity or intolerance to a human or humanized antibody or to BNT351 excipients

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Parts A and B - Occurrence of at least one adverse event (AE) | From dosing to 56 days post-dose
  Per part, by cohort/dose
Parts A and B - Occurrence of at least one serious AE (SAE) | From dosing through the end of study (up to a maximum of 279 days post-dose)
  Per part, by cohort/dose
Parts A and B (except for Cohort A1) - Occurrence of infusion-related reactions (IRRs) Grade ≥2 (graded based on National Cancer Institute Common Terminology Criteria for AEs [NCI CTCAE] version 5.0 as specified in the protocol) | From the start of IV dosing through 72 hours after the start of IV dosing
  Per part, by cohort/dose
Parts A and B - Occurrence of at least one solicited local reaction (pain/tenderness, erythema/redness, induration/swelling) at the investigational medicinal product administration site | From dosing through 7 days post-dose
  Per part, by cohort/dose
Parts A and B- Occurrence of at least one solicited systemic event (vomiting, diarrhea, headache, fatigue/malaise, myalgia/arthralgia, fever) | From dosing through 7 days post-dose
  Per part, by cohort/dose
Parts A and B- Assessment of area under the concentration-time curve of BNT351 | From pre-dose to last quantifiable timepoint (up to a maximum of 279 days post-dose)
  Per part, by cohort/dose
Parts A and B - Assessment of maximum concentration of BNT351 | From dosing through 7 days post-dose
  Per part, by cohort/dose
Part B - Occurrence of any acquired immunodeficiency syndrome (AIDS)-defining illness or opportunistic infection as defined in the protocol | From dosing up to the time of cART initiation (up to a maximum of 56 days post-dose)
Part B - Occurrence of absolute CD4+ T cell count <350 cells/µL or CD4+ T cell count <15% of total lymphocyte count | From dosing up to the time of cART initiation (up to a maximum of 56 days post-dose)
Part B - Change from baseline in HIV log10 plasma viral load prior to cART initiation | At 7, 14, 21, 28, 35, 42, 49, and 56 days post-dose
Part B - Maximum decrease from baseline in HIV log10 plasma viral load prior to cART initiation | From baseline up to the time of cART initiation (up to a maximum of 56 days post-dose)
Part B - Time from dosing to lowest viral load prior to cART initiation | From dosing up to the time of cART initiation (up to a maximum of 56 days post-dose)
Part B - Time from dosing to viral rebound defined as HIV-1 RNA viral load increase >0.75 log10 copies/mL from nadir (i.e., lowest HIV-1 RNA viral load from 7 days post-dose (Visit 3) and through pre-cART initiation) | From dosing up to the time of cART initiation (up to a maximum of 56 days post-dose)

SECONDARY OUTCOMES:
Parts A and B - Incidence of detectable BNT351 anti-drug antibodies in serum | From baseline until the end of study (up to a maximum of 279 days post-dose)
  Per part, by cohort/dose
Part B - Magnitude of cluster of differentiation 4 positive (CD4+) T cell counts | At dosing, 28 and 56 days post-dose or at time of cART initiation (up to a maximum of 56 days post-dose)
Parts B - Change from baseline in CD4+ T cell count | At 28 days post-dose and at time of cART initiation (up to a maximum of 56 days post-dose)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Response Person, Study Director — BioNTech SE

IPD SHARING:
Plan to Share IPD: No